CLINICAL TRIAL: NCT04583956
Title: A Multicenter Platform Trial of Putative Therapeutics for the Treatment of COVID-19 in Hospitalized Adults
Brief Title: ACTIV-5 / Big Effect Trial (BET-A) for the Treatment of COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-0013A
Record Dates: First submitted 2020-10-09; First posted 2020-10-12 (Actual); Results first posted 2022-12-19 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2021-09

CONDITIONS: COVID-19
Keywords: Adults; COVID-19; Multicenter; Platform; Putative; Therapeutics
MeSH Terms: conditions — COVID-19 | interventions — remdesivir; risankizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remdesivir + Placebo (Active Comparator): 200-mg intravenous (IV) remdesivir loading dose on Day 1, followed by a 100-mg once-daily IV maintenance dose up to a 10-day total course while hospitalized and 1200-mg IV risankizumab placebo infusion (300-mg x 4 vials) once on Day 1. N=100.
  Interventions: Other: Placebo; Drug: Remdesivir
- Remdesivir + Risankizumab (Experimental): 200-mg intravenous (IV) remdesivir loading dose on Day 1, followed by a 100-mg once-daily IV maintenance dose up to a 10-day total course while hospitalized and 1200-mg IV risankizumab infusion (300-mg x 4 vials) once on Day 1. N=100.
  Interventions: Drug: Remdesivir; Biological: Risankizumab

INTERVENTIONS:
Other: Placebo — Risankizumab placebo will be given at an equal volume at the same schedule.
  Arms: Remdesivir + Placebo
Drug: Remdesivir — Remdesivir is a single diastereomer monophosphoramidate prodrug for the intracellular delivery of a modified adenine nucleoside analog GS-441524.
Biological: Risankizumab — Risankizumab is a humanized immunoglobulin (Ig) G1 antagonistic monoclonal antibody (mAb) directed against the p19 subunit of the human cytokine interleukin-23. Risankizumab is formulated in a buffer of 4.4 mM disodium succinate hexahydrate/succinic acid, 225 mM sorbitol, 0.2 mg/mL polysorbate 20, and WFI in a 6R vial.
  Arms: Remdesivir + Risankizumab

SUMMARY:
This is a platform trial to conduct a series of randomized, double-blind, placebo-controlled trials using common assessments and endpoints in hospitalized adults diagnosed with Coronavirus Disease 2019 (COVID-19). Big Effect Trial (BET) is a proof-of-concept study with the intent of identifying promising treatments to enter a more definitive study. The study will be conducted in up to 70 domestic sites and 5 international sites. The study will compare different investigational therapeutic agents to a common control arm and determine which have relatively large effects. In order to maintain the double blind, each intervention will have a matched placebo. However, the control arm will be shared between interventions and may include participants receiving the matched placebo for a different intervention.

The goal is not to determine clear statistical significance for an intervention, but rather to determine which products have clinical data suggestive of efficacy and should be moved quickly into larger studies. Estimates produced from BET will provide an improved basis for designing the larger trial, in terms of sample size and endpoint selection. Products with little indication of efficacy will be dropped on the basis of interim evaluations. In addition, some interventions may be discontinued on the basis of interim futility or efficacy analyses.

One or more interventions may be started at any time. The number of interventions enrolling are programmatic decisions and will be based on the number of sites and the pace of enrollment. At the time of enrollment, subjects will be randomized to receive any one of the active arms they are eligible for or placebo. Approximately 200 (100 treatment and 100 shared placebo) subjects will be assigned to each arm entering the platform and a given site will generally have no more than 3 interventions at once.

The BET-A stage will evaluate the combination of remdesivir with risankizumab vs remdesivir with a risankizumab placebo. The primary objective is to evaluate the clinical efficacy of different investigational therapeutics relative to the control arm in adults hospitalized with COVID-19 according to clinical status (8-point ordinal scale) at Day 8.

DETAILED DESCRIPTION:
This is a platform trial to conduct a series of randomized, double-blind, placebo-controlled trials using common assessments and endpoints in hospitalized adults diagnosed with Coronavirus Disease 2019 (COVID-19). Big Effect Trial (BET) is a proof-of-concept study with the intent of identifying promising treatments to enter a more definitive study. The study will be conducted in up to 70 domestic sites and 5 international sites. The study will compare different investigational therapeutic agents to a common control arm and determine which have relatively large effects. In order to maintain the double blind, each intervention will have a matched placebo. However, the control arm will be shared between interventions and may include participants receiving the matched placebo for a different intervention.

The goal is not to determine clear statistical significance for an intervention, but rather to determine which products have clinical data suggestive of efficacy and should be moved quickly into larger studies. Estimates produced from BET will provide an improved basis for designing the larger trial, in terms of sample size and endpoint selection. Products with little indication of efficacy will be dropped on the basis of interim evaluations. In addition, some interventions may be discontinued on the basis of interim futility or efficacy analyses.

One or more interventions may be started at any time. The number of interventions enrolling are programmatic decisions and will be based on the number of sites and the pace of enrollment. At the time of enrollment, subjects will be randomized to receive any one of the active arms they are eligible for or placebo. Approximately 200 (100 treatment and 100 shared placebo) subjects will be assigned to each arm entering the platform and a given site will generally have no more than 3 interventions at once.

The BET-A stage will evaluate the combination of remdesivir with risankizumab vs remdesivir with a risankizumab placebo. Subjects will be assessed daily while hospitalized. Once subjects are discharged from the hospital, they will have a study visit at Days 8, 15, 22, 29, and 60 as an outpatient. The Day 8, Day 22 and Day 60 visits do not have laboratory tests or collection of samples and may be conducted by phone. All subjects will undergo a series of efficacy and safety laboratory assessments. Safety laboratory tests and blood (serum and plasma) research samples and oropharyngeal (OP) swabs will be obtained on Day 1 (prior to study product administration) and Days 3, 5, 8, and 11 while hospitalized. OP swabs (oropharyngeal swabs are preferred, but if these are not obtainable, saliva or nasopharyngeal or nasal swabs may be substituted) and blood research samples plus safety laboratory tests will be collected on Day 15 and 29 if the subject attends an in-person visit or is still hospitalized. However, if infection control considerations or other restrictions prevent the subject from returning to the clinic, Day 15 and 29 visits may be conducted by phone and only clinical data will be obtained.

The primary objective is to evaluate the clinical efficacy of different investigational therapeutics relative to the control arm in adults hospitalized with COVID-19 according to clinical status (8-point ordinal scale) at Day 8. The key secondary objectives are 1) to evaluate the clinical efficacy of different investigational therapeutics as assessed by time to recovery compared to the control arm, and 2) to evaluate the proportion of subjects alive and without respiratory failure through Day 29.

Contacts:

20-0013 Central Contact

Telephone: 1 (301) 7617948

Email: DMIDClinicalTrials@niaid.nih.gov

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to a hospital with symptoms suggestive of Coronavirus Disease 2019 (COVID-19) and requires ongoing medical care.
2. Subject (or legally authorized representative) provides informed consent prior to initiation of any study procedures.
3. Subject (or legally authorized representative) understands and agrees to comply with planned study procedures.
4. Male or non-pregnant female adult >/= 18 years of age at time of enrollment.
5. Illness of any duration and has laboratory-confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay (e.g., Nucleic Acid Amplification Test [NAAT], antigen test) in any respiratory specimen or saliva </=14 days prior to randomization.
6. Illness of any duration, and requiring, just prior to randomization, supplemental oxygen (any flow), mechanical ventilation or ECMO (ordinal score 5, 6, or 7).
7. Women of childbearing potential must agree to either abstinence or use at least one acceptable method of contraception from the time of screening through 5 months post study IP dosing.

   Note: Acceptable methods include barrier contraceptives (condoms or diaphragm) with spermicide, intrauterine devices (IUDs), hormonal contraceptives, oral contraceptive pills, and surgical sterilization.
8. Agrees not to participate in another blinded clinical trial (both pharmacologic and other types of interventions) for the treatment of COVID-19 through Day 29.

Exclusion Criteria:

1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the upper limit of normal.
2. Subjects with a low glomerular filtration rate (eGFR), specifically:

   1. Subjects with an a glomerular filtration rate (eGFR) 20-30 mL/min are excluded unless in the opinion of the principal investigator (PI), the potential benefit of participation outweighs the potential risk of study participation.
   2. All subjects with an a glomerular filtration rate (eGFR) <20 mL/min (including hemodialysis and hemofiltration) are excluded.
3. Pregnancy or breast feeding.
4. Anticipated discharge from the hospital or transfer to another hospital which is not a study site within 72 hours of enrollment.
5. Allergy to any study medication.
6. Received five or more doses of remdesivir prior to screening.
7. Received two or more doses of > 60 mg of prednisone or equivalent in the 7 days prior to screening.
8. Received small molecule tyrosine kinase inhibitors, including Janus kinase (JAK) inhibitors (e.g., baricitinib, ibrutinib, acalabrutinib, imatinib, gefitinib), in the 4 weeks prior to screening.
9. Received monoclonal antibodies targeting cytokines (e.g., tumor necrosis factor (TNF) inhibitors, anti-IL-1 [e.g., anakinra, canakinumab], anti-IL-6 [e.g., tocilizumab, sarilumab, sitlukimab]), or T-cells (e.g., abatacept) in the 4 weeks prior to screening.
10. Received monoclonal antibodies targeting B-cells (e.g., rituximab, and including any targeting multiple cell lines including B-cells) in the 3 months prior to screening.
11. Received Granulocyte-macrophage colony-stimulating factor (GM-CSF) agents (e.g., sargramostim) within 2 months prior to screening.
12. Received other immunosuppressants in the 4 weeks prior to screening and in the judgment of the investigator, the risk of immunosuppression with risankizumab is larger than the risk of Coronavirus Disease 2019 (COVID-19).
13. Received any live vaccine in the 4 weeks prior to screening.
14. Known active tuberculosis.
15. Known history of Human Immunodeficiency Virus (HIV), Hepatitis B (HBV) or untreated hepatitis C (HCV) infection.
16. History of pulmonary alveolar proteinosis (PAP).
17. Has a malignancy and currently receiving immunosuppressive chemotherapy, immunodeficiency, uncontrolled opportunistic infection, or uncontrolled cirrhosis.
18. Has a medical condition that could, in the judgment of the investigator, limit the interpretation and generalizability of trial results.
19. Positive test for influenza virus during the current illness (influenza testing is not required by protocol).
20. Previous participation in an ACTIV-5/Big Effect Trial (BET)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - The University of Arizona - Banner University Medical Center Tucson Campus - Tucson, Tucson, Arizona
  - Kern Medical Center, Bakersfield, California
  - Hoag Hospital Newport Beach, Newport Beach, California
  - Stanford University - Stanford Hospital and Clinics - Pediatrics - Infectious Diseases, Stanford, California
  - Penrose Hospital - Emergency Medicine, Colorado Springs, Colorado
  - St. Francis Medical Center, Colorado Springs, Colorado
  - St. Anthony Hospital, Lakewood, Colorado
  - St. Anthony Hospital North Health Campus, Westminster, Colorado
  - Nuvance Health Danbury Hospital - Infectious Disease, Danbury, Connecticut
  - Yale School of Medicine - The Anlyan Center for Medical Research & Education - Immunobiology, New Haven, Connecticut
  - Nuvance Health - Norwalk Hospital - Asthma Pulmonary and Critical Care Medicine, Norwalk, Connecticut
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - Cook County Health and Hospitals System - Ruth M Rothstein CORE Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Brigham and Women's Hospital - Infectious Diseases, Boston, Massachusetts
  - Boston Medical Center - Center for Infectious Diseases - Shapiro Center, Boston, Massachusetts
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota
  - University of Nebraska Medical Center- Infectious Diseases, Omaha, Nebraska
  - Englewood Hospital, Englewood, New Jersey
  - The State University of New York - University at Buffalo - Department of Medicine, Buffalo, New York
  - Mount Sinai School of Medicine - Medicine - Infectious Diseases, New York, New York
  - Nuvance Health - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Jacobi Medical Center, The Bronx, New York
  - Wake Forest Baptist Health - Infectious Diseases, Winston-Salem, North Carolina
  - University of Toledo Medical Center - Ruppert Clinic, Toledo, Ohio
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - Monument Health - Clinical Research, Rapid City, South Dakota
  - Hendrick Health - Hendrick Medical Center, Abilene, Texas
  - Baptist Hospitals of Southeast Texas Site, Beaumont, Texas
  - West Virginia University - Infectious Diseases Clinic, Morgantown, West Virginia

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were male and non-pregnant female adults =18 years of age or older and hospitalized with COVID-19. Participants were enrolled between 23OCT2020 and 13JUL2021.
Groups:
- Remdesivir + Risankizumab: 200-mg intravenous (IV) remdesivir loading dose on Day 1, followed by a 100-mg once-daily IV maintenance dose up to a 10-day total course while hospitalized and 1200-mg IV risankizumab infusion (300-mg x 4 vials) once on Day 1.
  Remdesivir: Remdesivir is a single diastereomer monophosphoramidate prodrug for the intracellular delivery of a modified adenine nucleoside analog GS-441524.
  Risankizumab: Risankizumab is a humanized immunoglobulin (Ig) G1 antagonistic monoclonal antibody (mAb) directed against the p19 subunit of the human cytokine interleukin-23. Risankizumab is formulated in a buffer of 4.4 mM disodium succinate hexahydrate/succinic acid, 225 mM sorbitol, 0.2 mg/mL polysorbate 20, and WFI in a 6R vial.
- Remdesivir + Placebo: 200-mg intravenous (IV) remdesivir loading dose on Day 1, followed by a 100-mg once-daily IV maintenance dose up to a 10-day total course while hospitalized and 1200-mg IV risankizumab placebo infusion (300-mg x 4 vials) once on Day 1.
  Placebo: Risankizumab placebo will be given at an equal volume at the same schedule.
  Remdesivir: Remdesivir is a single diastereomer monophosphoramidate prodrug for the intracellular delivery of a modified adenine nucleoside analog GS-441524.
Period: Overall Study
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Started | 104 | 110
Included in Modified Intention-to-treat (mITT) Population | 100 | 107
Completed | 83 | 85
Not Completed | 21 | 25
Not completed — Death | 9 | 11
Not completed — Lost to Follow-up | 7 | 9
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Randomized but not dosed | 2 | 3
Not completed — Withdrawal of consent before product administration | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intention-to-treat (ITT) population includes all participants who were enrolled and randomized.
Groups:
- Remdesivir + Risankizumab: 200-mg IV remdesivir loading dose on Day 1, followed by a 100-mg once-daily IV maintenance dose up to a 10-day total course while hospitalized and 1200-mg IV risankizumab infusion (300-mg x 4 vials) once on Day 1.
- Remdesivir + Placebo: 200-mg IV remdesivir loading dose on Day 1, followed by a 100-mg once-daily IV maintenance dose up to a 10-day total course while hospitalized and 1200-mg IV risankizumab placebo infusion (300-mg x 4 vials) once on Day 1.
- Total: Total of all reporting groups
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo | Total
Number analyzed (Participants) | 104 | 110 | 214
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 78 | 164
  >=65 years | 18 | 32 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (12.2) | 57.5 (13.1) | 56.0 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 52 | 88
  Male | 68 | 58 | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 20 | 43
  Not Hispanic or Latino | 81 | 89 | 170
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 6 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 28 | 53
  White | 59 | 67 | 126
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 8 | 20
Region of Enrollment [Number; unit: participants]
  United States | 104 | 110 | 214

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting Criteria for Each of the 8 Ordinal Scale Categories on Day 8
Description: The ordinal scale categories are defined as: 1) Not hospitalized, no new or increased limitations on activities; 2) Not hospitalized, but new or increased limitation on activities and/or requiring new or increased home oxygen, CPAP, or BiPAP; 3) Hospitalized, not requiring new or increased supplemental oxygen - no longer requires ongoing medical care; 4) Hospitalized, not requiring new or increased supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 5) Hospitalized, requiring new or increased supplemental oxygen; 6) Hospitalized, requiring new or increased non-invasive ventilation or high-flow oxygen devices; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 8) Death.
Time Frame: Day 8
Population: The modified intention-to-treat (mITT) population includes all randomized participants who received at least one dose of investigational product other than standard of care therapies, analyzed as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
Participants
  Not hospitalized, no new or increased limitations on activities | 15 | 21
  Not hosp., but new or incr. limit on activities and/or req. new or incr. home O2, CPAP, or BiPAP | 36 | 36
  Hospitalized, not req new or increased supplemental O2 - no longer req ongoing medical care | 0 | 0
  Hospitalized, not req new or increased supplemental O2 - req ongoing medical care | 6 | 3
  Hospitalized, requiring new or increased supplemental O2 | 17 | 16
  Hospitalized, requiring new or increased non-invasive ventilation or high-flow oxygen devices | 13 | 19
  Hospitalized, on invasive mechanical ventilation or ECMO | 11 | 9
  Death | 2 | 2
  Missing | 0 | 1
Statistical Analysis 1: Comparison: Remdesivir + Risankizumab vs Remdesivir + Placebo; Includes all ordinal score categories. Odds ratio of a better clinical status score, confidence interval, and p-value estimated from a proportional odds model adjusted for baseline steroid use and baseline ordinal score. Missing data imputed using multiple imputation (MI) for participants lost to follow-up before Day 8 while hospitalized, in hospice, long term acute care, or transferred to other hospital while participants lost to follow-up after discharge to home are assigned a score of 2; Test type: Superiority; p = 0.927, Proportional odds model; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.59 to 1.61] — Odds ratio above 1 favors Remdesivir plus Risankizumab

2. Secondary Outcome: Proportion of Participants Not Meeting Criteria for One of Two Ordinal Scale Categories Through Day 29
Description: Ordinal scale categories include 8) Death and 7) Hospitalized, on Invasive Mechanical Ventilation or Extracorporeal Membrane Oxygenation (ECMO). Mechanical ventilation-free survival was assessed through Day 29, defined as the proportion of participants who had not died nor were hospitalized on invasive mechanical ventilation or ECMO from Day 1 through Day 29. Results are reported as Kaplan Meier estimates.
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
Proportion of participants | 0.87 [0.78 to 0.92] | 0.88 [0.80 to 0.93]
Statistical Analysis 1: Comparison: Remdesivir + Risankizumab vs Remdesivir + Placebo; Odds ratio, confidence interval, and p-value estimated from a logistic regression model adjusted for baseline dexamethasone use, baseline ordinal score, age, and baseline C-Reactive Protein (CRP); Test type: Superiority; p = 0.829, Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.36 to 2.25] — Odds ratio greater than 1 favors Remdesivir plus Risankizumab

3. Secondary Outcome: Time to Sustained Recovery
Description: Day of sustained recovery is defined as the first day on which the participant satisfies 1 of the following 3 categories from the clinical status ordinal scale (and does not return to a score of = 4 up to and including Study Day 60): 1) Not hospitalized, no new or increased limitations on activities; 2) Not hospitalized, but new or increased limitation on activities and/or requiring new or increased home oxygen, CPAP, or BiPAP; 3) Hospitalized, not requiring new or increased supplemental oxygen - no longer requires ongoing medical care.
Time Frame: Day 1 through Day 60
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
days | 7.0 [5.0 to 8.0] | 6.0 [5.0 to 8.0]
Statistical Analysis 1: Comparison: Remdesivir + Risankizumab vs Remdesivir + Placebo; Hazard ratio, confidence interval, and p-value estimated from a Cox model adjusted for baseline steroid use and baseline ordinal score; Test type: Superiority; p = 0.399, Regression, Cox; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.84 to 1.56] — HR greater than 1 favors Remdesivir plus Risankizumab

4. Secondary Outcome: Number of Participants Meeting Criteria for Each of the 8 Ordinal Scale Categories on Day 15
Description: as for outcome 1
Time Frame: Day 15
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
Participants
  Not hospitalized, no new or increased limitations on activities | 31 | 37
  Not hosp., but new or incr. limit on activities and/or req. new or incr. home O2, CPAP, or BiPAP | 46 | 42
  Hospitalized, not req new or increased supplemental O2 - no longer req ongoing medical care | 0 | 0
  Hospitalized, not req new or increased supplemental O2 - req ongoing medical care | 1 | 2
  Hospitalized, requiring new or increased supplemental O2 | 10 | 10
  Hospitalized, requiring new or increased non-invasive ventilation or high-flow oxygen devices | 2 | 4
  Hospitalized, on invasive mechanical ventilation or ECMO | 4 | 9
  Death | 6 | 3
Statistical Analysis 1: Comparison: Remdesivir + Risankizumab vs Remdesivir + Placebo; Includes all ordinal score categories. Odds ratio of a better clinical status score, confidence interval, and p-value estimated from a proportional odds model adjusted for baseline steroid use and baseline ordinal score. Missing data imputed using last observation carried forward for those lost to follow-up before Day 15 while hospitalized, in hospice, long term acute care, or transferred to other hospital. Participants lost to follow-up before Day 15 after discharge are given a score of 2; Test type: Superiority; p = 0.910, Proportional odds model; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.62 to 1.71] — Odds ratio above 1 favors Remdesivir plus Risankizumab

5. Secondary Outcome: Number of Participants Meeting Criteria for Each of the 8 Ordinal Scale Categories on Day 29
Description: as for outcome 1
Time Frame: Day 29
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
Participants
  Not hospitalized, no new or increased limitations on activities | 46 | 50
  Not hosp., but new or incr. limit on activities and/or req. new or incr. home O2, CPAP, or BiPAP | 43 | 38
  Hospitalized, not req new or increased supplemental O2 - no longer req ongoing medical care | 0 | 0
  Hospitalized, not req new or increased supplemental O2 - req ongoing medical care | 0 | 1
  Hospitalized, requiring new or increased supplemental O2 | 0 | 3
  Hospitalized, requiring new or increased non-invasive ventilation or high-flow oxygen devices | 0 | 4
  Hospitalized, on invasive mechanical ventilation or ECMO | 4 | 4
  Death | 7 | 7
Statistical Analysis 1: Comparison: Remdesivir + Risankizumab vs Remdesivir + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.617, Proportional odds model; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.68 to 1.93] — Odds ratio above 1 favors Remdesivir plus Risankizumab

6. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP)
Description: Blood was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: The safety population includes all randomized participants who received at least one dose of investigational product other than standard of care therapies with available data at baseline and post baseline assessment time point, analyzed as treated.
Measure: Mean (Standard Deviation); unit: milligrams/liter (mg/L)
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
milligrams/liter (mg/L)
  Day 3: number analyzed (Participants) | 89 | 98
  Day 3 | -49.471 (68.217) | -37.344 (64.622)
  Day 5: number analyzed (Participants) | 66 | 72
  Day 5 | -64.340 (77.430) | -51.216 (80.230)
  Day 8: number analyzed (Participants) | 38 | 42
  Day 8 | -62.578 (82.042) | -58.094 (113.351)
  Day 11: number analyzed (Participants) | 17 | 26
  Day 11 | -17.365 (138.044) | -49.828 (143.271)
  Day 15: number analyzed (Participants) | 27 | 33
  Day 15 | -66.453 (76.258) | -58.816 (70.797)
  Day 29: number analyzed (Participants) | 28 | 31
  Day 29 | -77.527 (69.087) | -68.496 (74.662)

7. Secondary Outcome: Change From Baseline in Ferritin
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: micrograms/liter (ug/L)
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
micrograms/liter (ug/L)
  Day 3: number analyzed (Participants) | 88 | 95
  Day 3 | -187.123 (437.096) | -145.201 (562.150)
  Day 5: number analyzed (Participants) | 65 | 68
  Day 5 | -326.691 (610.633) | -37.041 (1956.100)
  Day 8: number analyzed (Participants) | 39 | 40
  Day 8 | -252.804 (754.932) | -236.725 (800.878)
  Day 11: number analyzed (Participants) | 17 | 26
  Day 11 | -90.829 (648.972) | -371.682 (628.049)
  Day 15: number analyzed (Participants) | 24 | 33
  Day 15 | -305.970 (941.210) | -317.063 (828.814)
  Day 29: number analyzed (Participants) | 29 | 31
  Day 29 | -520.237 (476.899) | -762.394 (1056.614)

8. Secondary Outcome: Change From Baseline in D-dimer
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ug/L fibrinogen equivalent units (FEU)
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
ug/L fibrinogen equivalent units (FEU)
  Day 3: number analyzed (Participants) | 87 | 96
  Day 3 | -1642.4 (12710.1) | -38.8 (3315.6)
  Day 5: number analyzed (Participants) | 64 | 68
  Day 5 | -914.1 (21635.7) | -129.3 (4104.4)
  Day 8: number analyzed (Participants) | 39 | 37
  Day 8 | -4124.4 (23690.0) | -38.9 (19399.8)
  Day 11: number analyzed (Participants) | 18 | 26
  Day 11 | -10670.7 (34100.4) | -741.2 (5094.4)
  Day 15: number analyzed (Participants) | 26 | 35
  Day 15 | -8990.9 (28348.8) | 907.1 (8625.0)
  Day 29: number analyzed (Participants) | 24 | 29
  Day 29 | -6516.8 (20705.8) | -471.8 (2401.0)

9. Secondary Outcome: Change From Baseline in Fibrinogen
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: milligrams/deciliter (mg/dL)
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
milligrams/deciliter (mg/dL)
  Day 3: number analyzed (Participants) | 82 | 87
  Day 3 | -89.7 (124.9) | -78.6 (109.6)
  Day 5: number analyzed (Participants) | 62 | 62
  Day 5 | -109.0 (169.3) | -108.8 (165.1)
  Day 8: number analyzed (Participants) | 36 | 34
  Day 8 | -100.5 (218.2) | -121.0 (225.5)
  Day 11: number analyzed (Participants) | 18 | 23
  Day 11 | 61.1 (319.3) | -33.2 (282.7)
  Day 15: number analyzed (Participants) | 22 | 31
  Day 15 | -37.6 (235.1) | -26.3 (181.6)
  Day 29: number analyzed (Participants) | 22 | 27
  Day 29 | -99.3 (208.1) | -102.0 (185.6)

10. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT)
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
U/L
  Day 3: number analyzed (Participants) | 98 | 103
  Day 3 | 6.1 (25.8) | 9.6 (43.5)
  Day 5: number analyzed (Participants) | 72 | 77
  Day 5 | 9.4 (34.7) | 64.0 (290.4)
  Day 8: number analyzed (Participants) | 43 | 43
  Day 8 | 6.1 (48.3) | 33.9 (168.1)
  Day 11: number analyzed (Participants) | 20 | 27
  Day 11 | 5.3 (55.7) | 21.5 (117.7)
  Day 15: number analyzed (Participants) | 31 | 34
  Day 15 | 7.6 (45.9) | -3.3 (55.3)
  Day 29: number analyzed (Participants) | 34 | 34
  Day 29 | -0.1 (31.6) | -19.3 (62.1)

11. Secondary Outcome: Change From Baseline in Aspartate Transaminase (AST)
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
U/L
  Day 3: number analyzed (Participants) | 98 | 103
  Day 3 | -1.4 (39.9) | -5.0 (46.4)
  Day 5: number analyzed (Participants) | 72 | 77
  Day 5 | -8.4 (36.6) | 44.2 (432.3)
  Day 8: number analyzed (Participants) | 43 | 43
  Day 8 | -16.7 (37.6) | 34.9 (404.0)
  Day 11: number analyzed (Participants) | 20 | 27
  Day 11 | -8.9 (45.1) | 39.4 (318.0)
  Day 15: number analyzed (Participants) | 30 | 34
  Day 15 | -13.8 (34.6) | -16.9 (33.0)
  Day 29: number analyzed (Participants) | 34 | 34
  Day 29 | -13.1 (22.4) | -28.2 (37.3)

12. Secondary Outcome: Change From Baseline in Hemoglobin
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
g/dL
  Day 3: number analyzed (Participants) | 97 | 103
  Day 3 | -0.199 (0.785) | -0.035 (0.893)
  Day 5: number analyzed (Participants) | 73 | 77
  Day 5 | -0.485 (1.142) | -0.074 (1.202)
  Day 8: number analyzed (Participants) | 41 | 43
  Day 8 | -0.461 (1.434) | -0.323 (1.460)
  Day 11: number analyzed (Participants) | 19 | 28
  Day 11 | -1.079 (1.997) | -0.714 (1.722)
  Day 15: number analyzed (Participants) | 30 | 37
  Day 15 | -0.817 (1.702) | -0.805 (1.929)
  Day 29: number analyzed (Participants) | 33 | 33
  Day 29 | -0.524 (1.989) | -0.642 (1.867)

13. Secondary Outcome: Change From Baseline in Creatinine
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
mg/dL
  Day 3: number analyzed (Participants) | 98 | 104
  Day 3 | 0.000 (0.332) | -0.858 (8.777)
  Day 5: number analyzed (Participants) | 74 | 78
  Day 5 | -0.041 (0.306) | -1.091 (10.138)
  Day 8: number analyzed (Participants) | 43 | 43
  Day 8 | -0.023 (0.281) | -1.993 (13.677)
  Day 11: number analyzed (Participants) | 20 | 28
  Day 11 | -0.127 (0.371) | -3.044 (16.911)
  Day 15: number analyzed (Participants) | 31 | 35
  Day 15 | -0.096 (0.347) | 0.362 (1.172)
  Day 29: number analyzed (Participants) | 34 | 34
  Day 29 | -0.023 (0.249) | 0.211 (1.148)

14. Secondary Outcome: Change From Baseline in International Normalized Ratio (INR)
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
Ratio
  Day 3: number analyzed (Participants) | 88 | 98
  Day 3 | 0.063 (0.174) | 0.069 (0.257)
  Day 5: number analyzed (Participants) | 65 | 68
  Day 5 | 0.103 (0.257) | 0.174 (0.682)
  Day 8: number analyzed (Participants) | 36 | 38
  Day 8 | 0.038 (0.206) | 0.277 (1.580)
  Day 11: number analyzed (Participants) | 19 | 26
  Day 11 | 0.137 (0.525) | 0.015 (0.249)
  Day 15: number analyzed (Participants) | 26 | 34
  Day 15 | -0.092 (0.238) | -0.077 (0.164)
  Day 29: number analyzed (Participants) | 27 | 31
  Day 29 | -0.129 (0.185) | -0.075 (0.141)

15. Secondary Outcome: Change From Baseline in Platelets
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
10^9 cells/L
  Day 3: number analyzed (Participants) | 97 | 103
  Day 3 | 59.49 (48.59) | 50.45 (60.91)
  Day 5: number analyzed (Participants) | 73 | 77
  Day 5 | 81.22 (65.53) | 76.17 (80.11)
  Day 8: number analyzed (Participants) | 40 | 43
  Day 8 | 96.73 (106.11) | 71.59 (139.53)
  Day 11: number analyzed (Participants) | 19 | 28
  Day 11 | 54.95 (109.38) | -1.68 (117.94)
  Day 15: number analyzed (Participants) | 30 | 37
  Day 15 | -16.90 (110.76) | -24.19 (120.42)
  Day 29: number analyzed (Participants) | 33 | 33
  Day 29 | 27.42 (128.22) | 45.97 (111.20)

16. Secondary Outcome: Change From Baseline in Bilirubin
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
mg/dL
  Day 3: number analyzed (Participants) | 97 | 102
  Day 3 | -0.033 (0.201) | -0.024 (0.152)
  Day 5: number analyzed (Participants) | 72 | 76
  Day 5 | -0.020 (0.267) | 0.026 (0.249)
  Day 8: number analyzed (Participants) | 43 | 43
  Day 8 | 0.016 (0.336) | 0.076 (0.343)
  Day 11: number analyzed (Participants) | 19 | 27
  Day 11 | 0.153 (0.467) | 0.148 (0.581)
  Day 15: number analyzed (Participants) | 30 | 34
  Day 15 | 0.157 (0.494) | 0.131 (0.430)
  Day 29: number analyzed (Participants) | 33 | 34
  Day 29 | -0.033 (0.291) | -0.091 (0.223)

17. Secondary Outcome: Change From Baseline in White Blood Cell (WBC)
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
10^9 cells/L
  Day 3: number analyzed (Participants) | 97 | 103
  Day 3 | 1.672 (3.589) | 1.432 (3.453)
  Day 5: number analyzed (Participants) | 73 | 77
  Day 5 | 2.484 (4.053) | 2.437 (4.231)
  Day 8: number analyzed (Participants) | 41 | 43
  Day 8 | 3.726 (3.781) | 5.298 (6.390)
  Day 11: number analyzed (Participants) | 19 | 28
  Day 11 | 4.852 (6.784) | 4.545 (7.772)
  Day 15: number analyzed (Participants) | 30 | 37
  Day 15 | 1.770 (5.869) | 1.663 (5.882)
  Day 29: number analyzed (Participants) | 32 | 33
  Day 29 | -0.801 (4.355) | -2.016 (4.645)

18. Secondary Outcome: Change From Baseline in Neutrophils
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
10^9 cells/L
  Day 3: number analyzed (Participants) | 80 | 85
  Day 3 | 1.0297 (2.6919) | 0.9628 (3.0963)
  Day 5: number analyzed (Participants) | 56 | 62
  Day 5 | 1.1050 (2.6733) | 1.3373 (3.3580)
  Day 8: number analyzed (Participants) | 31 | 35
  Day 8 | 2.8066 (3.1523) | 4.1114 (5.5771)
  Day 11: number analyzed (Participants) | 13 | 23
  Day 11 | 4.0192 (5.5099) | 2.4704 (4.7446)
  Day 15: number analyzed (Participants) | 25 | 30
  Day 15 | -0.5410 (2.9101) | 0.1833 (3.5524)
  Day 29: number analyzed (Participants) | 22 | 25
  Day 29 | -1.8493 (3.3028) | -2.6216 (3.8118)

19. Secondary Outcome: Change From Baseline in Eosinophils
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
10^9 cells/L
  Day 3: number analyzed (Participants) | 71 | 79
  Day 3 | 0.0009 (0.0350) | 0.0062 (0.0557)
  Day 5: number analyzed (Participants) | 51 | 59
  Day 5 | 0.0297 (0.0615) | 0.0221 (0.0699)
  Day 8: number analyzed (Participants) | 27 | 32
  Day 8 | 0.0810 (0.0969) | 0.0259 (0.0717)
  Day 11: number analyzed (Participants) | 11 | 22
  Day 11 | 0.1282 (0.1387) | 0.0814 (0.0953)
  Day 15: number analyzed (Participants) | 25 | 28
  Day 15 | 0.0924 (0.0902) | 0.1761 (0.1577)
  Day 29: number analyzed (Participants) | 22 | 24
  Day 29 | 0.1256 (0.0955) | 0.3421 (0.3291)

20. Secondary Outcome: Change From Baseline in Basophils
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
10^9 cells/L
  Day 3: number analyzed (Participants) | 72 | 81
  Day 3 | 0.0101 (0.0561) | 0.0052 (0.0286)
  Day 5: number analyzed (Participants) | 49 | 57
  Day 5 | 0.0038 (0.0315) | 0.0039 (0.0275)
  Day 8: number analyzed (Participants) | 27 | 31
  Day 8 | 0.0455 (0.2018) | 0.0061 (0.0308)
  Day 11: number analyzed (Participants) | 11 | 22
  Day 11 | 0.0291 (0.0288) | 0.0123 (0.0357)
  Day 15: number analyzed (Participants) | 25 | 28
  Day 15 | 0.0202 (0.0348) | 0.0254 (0.0307)
  Day 29: number analyzed (Participants) | 22 | 24
  Day 29 | 0.0262 (0.0343) | 0.0425 (0.0387)

21. Secondary Outcome: Change From Baseline in Lymphocytes
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
10^9 cells/L
  Day 3: number analyzed (Participants) | 80 | 84
  Day 3 | 0.2788 (0.4560) | 0.3009 (0.5398)
  Day 5: number analyzed (Participants) | 56 | 61
  Day 5 | 0.4256 (0.6067) | 0.4233 (0.7375)
  Day 8: number analyzed (Participants) | 30 | 33
  Day 8 | 0.3956 (0.6478) | 0.2612 (0.6765)
  Day 11: number analyzed (Participants) | 13 | 22
  Day 11 | 0.4431 (0.5793) | 0.2932 (0.6446)
  Day 15: number analyzed (Participants) | 25 | 28
  Day 15 | 0.7937 (0.6577) | 0.6096 (0.7233)
  Day 29: number analyzed (Participants) | 22 | 24
  Day 29 | 0.8309 (0.5085) | 0.7879 (0.5810)

22. Secondary Outcome: Change From Baseline in Monocytes
Description: as for outcome 6
Time Frame: Days 1, 3, 5, 8, 11, 15, 29
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
10^9 cells/L
  Day 3: number analyzed (Participants) | 79 | 84
  Day 3 | 0.1697 (0.3201) | 0.1023 (0.5020)
  Day 5: number analyzed (Participants) | 55 | 61
  Day 5 | 0.2023 (0.3254) | 0.1318 (0.5708)
  Day 8: number analyzed (Participants) | 28 | 34
  Day 8 | 0.3398 (0.4427) | 0.1135 (0.7707)
  Day 11: number analyzed (Participants) | 12 | 23
  Day 11 | 0.2450 (0.2887) | 0.1835 (0.8518)
  Day 15: number analyzed (Participants) | 24 | 29
  Day 15 | 0.1694 (0.3182) | 0.1407 (0.6706)
  Day 29: number analyzed (Participants) | 22 | 25
  Day 29 | -0.0175 (0.2896) | -0.0232 (0.7208)

23. Secondary Outcome: Number of Participants Reporting Grade 3 and 4 Clinical and/or Laboratory Adverse Events (AEs)
Description: Grade 3 AEs are defined as events that interrupt usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. Severe events are usually incapacitating. Grade 4 AEs are defined as events that are potentially life threatening.
Time Frame: Day 1 through Day 60
Population: The safety population includes all randomized participants who received at least one dose of investigational product other than standard of care therapies, analyzed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
Participants | 42 | 46

24. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: An SAE is defined as an AE or suspected adverse reaction that is considered serious if, in the view of either the investigator or the sponsor, it results in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Day 1 through Day 60
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
Participants | 24 | 26

25. Secondary Outcome: Number of Participants Who Discontinued or Temporarily Suspended Study Treatment
Description: Discontinuation or temporary suspension of study product is defined as any episode of early discontinuation or interruption of study product administration.
Time Frame: Day 1 through Day 29
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
Participants | 1 | 0

26. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization is defined first as the total number of days hospitalized for COVID-19, including readmissions for COVID-19-related reasons. It is also calculated as the total number of days hospitalized, including any readmissions for any reason.
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
days
  Hospitalized for COVID-19 | 6.0 [4.0 to 11.5] | 6.0 [4.0 to 13.0]
  Hospitalized for Any Reason | 6.0 [4.0 to 11.5] | 6.0 [4.0 to 14.0]

27. Secondary Outcome: Days of New Invasive Mechanical Ventilation / Extracorporeal Membrane Oxygenation (ECMO) Use
Description: Duration of new invasive mechanical ventilation/ECMO use was measured in days among participants not on invasive ventilation/ECMO at baseline who progressed to invasive ventilation/ECMO or died.
Time Frame: Day 1 through Day 29
Population: The modified intention-to-treat (mITT) population includes all randomized participants who received at least one dose of investigational product other than standard of care therapies, analyzed as randomized. Only participants not on invasive ventilation/ECMO at baseline were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 97 | 104
days | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

28. Secondary Outcome: Days of Non-invasive Ventilation/High Flow Oxygen Use
Description: Duration of non-invasive ventilation or high flow oxygen use was measured in days among participants who required non-invasive ventilation/high flow oxygen, invasive ventilation/ECMO or died.
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
days | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 7.0]

29. Secondary Outcome: Days of New Non-invasive Ventilation/High Flow Oxygen Use
Description: Duration of new non-invasive ventilation or high flow oxygen use was measured in days among participants not on non-invasive ventilation/high flow oxygen at baseline who progressed to non-invasive ventilation/high flow oxygen, invasive ventilation/ECMO or died.
Time Frame: Day 1 through Day 29
Population: The modified intention-to-treat (mITT) population includes all randomized participants who received at least one dose of investigational product other than standard of care therapies, analyzed as randomized. Only participants in the hospitalized requiring new or increased supplemental oxygen ordinal scale or below at baseline were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 69 | 79
days | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 1.0]

30. Secondary Outcome: Number of Participants With New Invasive Mechanical Ventilation / Extracorporeal Membrane Oxygenation (ECMO) Use
Description: New Invasive Mechanical Ventilation / Extracorporeal Membrane Oxygenation (ECMO) Use is defined as participants not on invasive ventilation/ECMO at baseline who progressed to invasive ventilation/ECMO or died during the study.
Time Frame: Day 1 through Day 29
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 97 | 104
Participants | 12 | 12

31. Secondary Outcome: Number of Participants With New Non-invasive Ventilation/High Flow Oxygen Use
Description: New Non-invasive Ventilation/High Flow Oxygen Use is defined as participants in the hospitalized requiring new or increased supplemental oxygen ordinal scale or below at baseline who progressed to non-invasive ventilation/high flow oxygen, invasive ventilation/ECMO or died during the study.
Time Frame: Day 1 through Day 29
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 69 | 79
Participants | 10 | 20

32. Secondary Outcome: Mean Change in Ordinal Scale
Description: The ordinal scale categories are defined as: 1) Not hospitalized, no new or increased limitations on activities;2) Not hospitalized, but new or increased limitation on activities and/or requiring new or increased home oxygen, CPAP, or BiPAP; 3) Hospitalized, not requiring new or increased supplemental oxygen - no longer requires ongoing medical care; 4)Hospitalized, not requiring new or increased supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 5) Hospitalized, requiring new or increased supplemental oxygen; 6) Hospitalized, requiring new or increased non-invasive ventilation or high-flow oxygen devices; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 8) Death. A positive change indicates a worsening and a negative change is an improvement.
Time Frame: Day 1, 3, 5, 11, 15, 22, 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
units on a scale
  Day 3 | 0.0 (0.5) | 0.0 (0.4)
  Day 5 | -0.5 (1.3) | -0.4 (1.2)
  Day 8 | -1.7 (1.9) | -1.7 (2.0)
  Day 11 | -2.2 (1.9) | -2.1 (2.0)
  Day 15 | -2.7 (1.9) | -2.6 (1.9)
  Day 22 | -3.1 (1.9) | -2.8 (1.8)
  Day 29 | -3.2 (1.9) | -2.9 (1.9)

33. Secondary Outcome: Proportion of Participants Not Meeting Criteria for One of Two Ordinal Scale Categories at Day 29
Description: Ordinal scale categories include 8) Death and 7) Hospitalized, on Invasive Mechanical Ventilation or Extracorporeal Membrane Oxygenation (ECMO). Defined as the proportion of participants who were alive and were not hospitalized on invasive mechanical ventilation or ECMO at the Day 29 visit.
Time Frame: Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
Proportion of participants | 0.89 [0.81 to 0.94] | 0.90 [0.83 to 0.95]

34. Secondary Outcome: 14-day Participant Mortality
Description: The mortality rate was determined as the proportion of participants who died by study Day 15. The proportions reported are Kaplan-Meier estimates.
Time Frame: Day 1 through Day 15
Population: The safety population includes all randomized participants who received at least one dose of investigational product other than standard of care therapies, classified by their actual treatment assignment.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
Proportion of participants | 0.06 [0.03 to 0.13] | 0.03 [0.01 to 0.08]

35. Secondary Outcome: 28-day Participant Mortality
Description: The mortality rate was determined as the proportion of participants who died by study Day 29. The proportions reported are Kaplan-Meier estimates.
Time Frame: Day 1 through Day 29
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
Proportion of participants | 0.07 [0.04 to 0.15] | 0.08 [0.04 to 0.15]

36. Secondary Outcome: 59-day Participant Mortality
Description: The mortality rate was determined as the proportion of participants who died by study Day 60. The proportions reported are Kaplan-Meier estimates.
Time Frame: Day 1 through Day 60
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
Proportion of participants | 0.09 [0.05 to 0.17] | 0.11 [0.06 to 0.19]

37. Secondary Outcome: Days of Supplemental Oxygen Use
Description: Duration of supplemental oxygen use was measured in days among participants who required any supplemental oxygen, non-invasive ventilation/high flow oxygen, invasive ventilation/ECMO or died.
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
days | 11.0 [4.0 to 28.0] | 11.0 [5.0 to 28.0]

38. Secondary Outcome: Time to an Improvement of One Category From Baseline Using an Ordinal Scale
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Not hospitalized, no new or increased limitations on activities; 2) Not hospitalized, but new or increased limitation on activities and/or requiring new or increased home oxygen, CPAP, or BiPAP; 3) Hospitalized, not requiring new or increased supplemental oxygen - no longer requires ongoing medical care; 4) Hospitalized, not requiring new or increased supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 5) Hospitalized, requiring new or increased supplemental oxygen; 6) Hospitalized, requiring new or increased non-invasive ventilation or high-flow oxygen devices; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 8) Death.
Time Frame: Day 1 through Day 60
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
days | 6.0 [6.0 to 7.0] | 7.0 [6.0 to 8.0]
Statistical Analysis 1: Comparison: Remdesivir + Risankizumab vs Remdesivir + Placebo; Hazard ratio (HR), confidence interval, and p-value estimated from a Cox model adjusted for baseline steroid use and baseline ordinal score; Test type: Superiority; p = 0.550, Regression, Cox; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.82 to 1.46] — HR greater than 1 favors Remdesivir plus Risankizumab

39. Secondary Outcome: Time to an Improvement of Two Categories From Baseline Using an Ordinal Scale
Description: as for outcome 38
Time Frame: Day 1 through Day 60
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
days | 12.0 [10.0 to 13.0] | 13.0 [9.0 to 13.0]
Statistical Analysis 1: Comparison: Remdesivir + Risankizumab vs Remdesivir + Placebo; [analysis description as in outcome 38, analysis 1]; Test type: Superiority; p = 0.523, Regression, Cox; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.82 to 1.48] — HR greater than 1 favors Remdesivir plus Risankizumab

40. Secondary Outcome: Time to Death
Description: The time death from study Day 1 to study Day 29, measured in days. The times reported are Kaplan-Meier estimates.
Time Frame: Day 1 through Day 29
Population: as for outcome 34
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
days | NA [NA to NA] — Median, lower and upper confidence intervals were not reached due to insufficient number of participants with events (deaths). | NA [NA to NA] — Median, lower and upper confidence intervals were not reached due to insufficient number of participants with events (deaths).

41. Secondary Outcome: Days of Invasive Mechanical Ventilation / Extracorporeal Membrane Oxygenation (ECMO) Use
Description: Duration of invasive ventilation/ECMO was measured in days among participants who required invasive ventilation or died.
Time Frame: Day 1 through Day 29
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
Number analyzed (Participants) | 100 | 107
days | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

ADVERSE EVENTS:
Time Frame: Grade 3 and 4 serious and non-serious adverse events were collected for 60 days after the first dose. Laboratory values were systematically assessed at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29.
Description: Given the nature of severity of the underlying illness, participants were expected to have many symptoms and abnormalities in vital signs and laboratory values. Per protocol, AEs specified to be captured in this trial included all Grade 3 and 4 AEs and any Grade 2 or higher, suspected drug-related hypersensitivity reactions. All cause mortality was calculated for the ITT population, while SAEs and AEs reflect the as treated population.
Groups:
- Remdesivir + Risankizumab: 200-mg intravenous (IV) remdesivir loading dose on Day 1, followed by a 100-mg once-daily IV maintenance dose up to a 10-day total course while hospitalized and 1200-mg IV risankizumab infusion (300-mg x 4 vials) once on Day 1.
- Remdesivir + Placebo: 200-mg intravenous (IV) remdesivir loading dose on Day 1, followed by a 100-mg once-daily IV maintenance dose up to a 10-day total course while hospitalized and 1200-mg IV risankizumab placebo infusion (300-mg x 4 vials) once on Day 1.
Arm/Group | Remdesivir + Risankizumab | Remdesivir + Placebo
All-Cause Mortality (participants affected / at risk) | 9/104 | 11/110
Serious Adverse Events (participants affected / at risk) | 24/100 | 26/107
Other Adverse Events (participants affected / at risk) | 24/100 | 22/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remdesivir + Risankizumab (N=100) | Remdesivir + Placebo (N=107)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Incarcerated hernia (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Obstruction (General disorders) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 3 (4)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 3 (3) | 4 (5)
Chillblains (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Body temperature decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3)
Renal Failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 8 (9)
Extubation (Surgical and medical procedures) | 1 (1) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remdesivir + Risankizumab (N=100) | Remdesivir + Placebo (N=107)
Glomerular filtration rate decreased (Investigations) | 8 (10) | 5 (6)
Lymphocyte count decreased (Investigations) | 6 (8) | 6 (6)
Oxygen saturation decreased (Investigations) | 5 (5) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 6 (6)
Hypertension (Vascular disorders) | 4 (4) | 10 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT04583956/Prot_004.pdf
  • Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT04583956/SAP_003.pdf
  • Informed Consent Form (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT04583956/ICF_001.pdf